CLINICAL TRIAL: NCT04585659
Title: Qigong for Multiple Sclerosis: A Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Natural Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 102015
Record Dates: First submitted 2020-09-02; First posted 2020-10-14 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-09

CONDITIONS: Multiple Sclerosis
Keywords: Qigong; Pragmatic Design; Gait; Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Qigong

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Qigong Intervention (Experimental): 60-90 minute community qigong classes, once per week plus at least 10 minutes of home practice
  Interventions: Other: Qigong
- Wait-List Control (No Intervention): Participants asked not to do any qigong, yoga or taichi for 10 weeks. Participants have the option to cross-over to the experimental arm after 10 weeks of no intervention.

INTERVENTIONS:
Other: Qigong — Mind-body movement art that includes specific movements, breath exercises, stretching and meditation.
  Other Names: Qi-gong
  Arms: Qigong Intervention

SUMMARY:
This feasibility study explores a community-based qigong intervention for people with multiple sclerosis (MS). The primary aim is to assess the feasibility of weekly community qigong classes for people with MS. The secondary aim is to explore the effects of qigong on balance, gait, mood, fatigue, and quality of life.

DETAILED DESCRIPTION:
Qigong, a traditional Chinese mind-body exercise, has been shown to improve balance and gait in several neurological conditions; however, community-delivered qigong has never been assessed for people with multiple sclerosis (MS). We assessed the feasibility of community qigong classes for people with MS and explored outcomes of balance, gait, and quality of life (QOL).

Twenty adults with MS were randomly assigned to 10 weeks of community qigong classes or wait-list control. Feasibility criteria included recruitment, retention, adherence, and ability to participate in qigong movements. Secondary outcome measures included physical tests of mobility, gait and balance, and participant-reported mobility, depression, anxiety, fatigue, and QOL.

Because this is a small feasibility study, the data collected are meant to be hypothesis-generating. Any clinically meaningful trends toward improvement will justify further exploration of qigong for MS in a larger clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Living in the Portland Metropolitan Area
* Self-reported diagnosis of multiple sclerosis (MS - any type)
* Demonstrated ability to walk 50 feet without assistance
* Stable on disease-modifying or balance medications three months prior to baseline

Exclusion Criteria:

* Pregnant or nursing
* Participated in qigong, tai chi, or yoga (>1 month) within six months prior to baseline
* Had an MS relapse within 30 days prior to baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-03-16 (Actual); Study Completion 2018-03-16 (Actual)

PRIMARY OUTCOMES:
Feasibility Outcome 1: Number of participants recruited for the study | 8 months
  Ability to recruit and enroll 20 participants with multiple sclerosis (MS) within 8 months.
Feasibility Outcome 2: Number of participants retained in the study | 10 weeks
  Goal to retain 80 percent of participants in the trial.
Feasibility Outcome 3: Percent able to participate in qigong classes | 10 weeks
  Participation based on participants' subjective report at week 1, 2, 7 phone check-ins and exit survey. Participants select from the following options: full participation, partial, a little, or none.
Feasibility Outcome 4: Percent attendance in qigong classes | 10 weeks
  Class attendance measured by self-report in exit survey and tracked by qigong instructor, with the goal of 70 percent attendance in class.

SECONDARY OUTCOMES:
Clinical Measure 1: Walking speed assessed by the Timed-25-Foot-Walk Test | Baseline and 10 weeks
  The Timed-25-Foot-Walk (T25FW) reliably measures walking ability for people with MS, and has a high test-retest reliability (intraclass correlation coefficient (ICC) of 0.99). The test is administered and rated by a trained examiner, and consists of having the participant walk a 25-foot long course as quickly as safely possible while being timed. Once the subject reaches the end-point, he/she is asked to turn around and walk back through the course, also while being timed. The score is an average of the time needed to complete each of the two trials. Lower scores indicate faster walking ability.
Clinical Measure 2: Mobility, balance and walking ability assessed by the Timed-Up-and-Go Test | Baseline and 10 weeks
  The Timed-Up-and-Go tests muscle function and mobility, predicts safe walking ability, and correlates with other mobility tests (r=0.81 correlation with Berg Balance Scale, r=-0.61 for gait speed). The test begins with the participant sitting in an armchair with his/her back resting on the back of the chair and arms resting on the arms of the chair. The participant is then asked to stand up and walk 3 m at a comfortable and safe speed, turn around, walk back and return to a seated position. The time that it takes to complete this exercise is then recorded. Lower scores indicate faster walking ability.
Clinical Measure 3: Multidirectional mobility assessed by the Four-Square-Step-Test | Baseline and 10 weeks
  The Four-Square-Step-Test is a validated measure of multi-directional mobility for MS, with high interrater (ICC=0.99) and retest reliability (ICC=0.98). The test measures a person's ability to step over objects in four directions. We created 4 3-ft boxes on the floor using colored masking tape. Participants are asked to step from the first box forward to the second, then right to square 3, back to square 4, and left to square 1, and then go back in the opposite order (4 to 3 to 2 to 1) while being timed. The participant is allowed practice this sequence before being timed. The test is repeated twice, with the best time taken as the score. Lower scores indicate greater multi-directional mobility.
Clinical Measure 4: Physical and psychological well-being assessed by the Multiple Sclerosis Impact Scale (MSIS-29) | Baseline and 10 weeks
  The Multiple Sclerosis Impact Scale (MSIS-29) is a validated core outcome measure that allows people with multiple sclerosis (MS) to self-assess the impact of MS on their physical and psychological well-being. This scale is commonly used to assess quality of life in studies of exercise and MS. The MSIS-29 was developed in 2000 as a patient-administered survey for MS, and includes 20 questions on physical impacts and 9 questions on psychological impacts of MS.55 The MSIS scales have good variability, small floor-to-ceiling effects, high internal consistency (Cronbach's alpha < 0.91), and high test-retest reliability (intraclass correlation > 0.87). Scores are adjusted to a 0 (min) to100 (max) scale. Higher scores indicate a worsening or more severe impact of MS on a person's physical and/or psychological condition.
Clinical Measure 5: Impact of multiple sclerosis on walking ability assessed by the Multiple Sclerosis Walking Scale (MSWS-12) | Baseline and 10 weeks
  The MS Walking Scale is a 12-question self-reported measure of impact of MS on walking ability. The test has good test-retest reliability (intraclass correlation > 0.78), and high internal consistency, criterion validity, and reliability (> 0.94). We included this measure to complement the physical tests on balance and gait. Scores are adjusted to a 0-100 scale. Higher scores indicate a greater impact of MS on walking ability (i.e., more difficulty walking).
Clinical Measure 6: Fatigue assessed by the Modified Fatigue Impact Scale Short Version (MFIS-5) | Baseline and 10 weeks
  The Modified Fatigue Impact Scale (MFIS) has been recommended by the ICM as a measure of energy and drive. The measure assesses physical, cognitive and psychosocial aspects of fatigue, and has a high internal consistency (Cronbach's alpha of 0.80). The 5-item version takes 2 minutes to complete, has an adequate test-retest reliability (r=0.76), and has been shown to capture meaningful changes in fatigue. Scores range from 0-20. Higher scores indicate higher levels of fatigue.
Clinical Measure 7: Health-related quality of life assessed by the Patient Reported Outcomes Measurement Information System global heath (mental and physical, v1.1) | Baseline and 10 weeks
  Patient Reported Outcomes Measurement Information System (PROMIS) are patient reported outcome surveys developed by the National Institutes for Health. The minimum raw score is 4, and maximum is 20. Raw scores are converted to standardized T-scores relative to a population mean of 50 and SD of 10 (T-scores range from 16.2 (minimum) to 67.7 (maximum) for physical measures, and 21.2-67.6 for mental). Higher T-scores represent higher levels of global health. Scores are calibrated against the general population.
Clinical Measure 8: Health-related quality of life assessed by the Patient Reported Outcomes Measurement Information System physical function (v1.2) | Baseline and 10 weeks
  Patient Reported Outcomes Measurement Information System (PROMIS) are patient reported outcome surveys developed by the National Institutes for Health. This test is a computer adaptive test. Scores are represented as standardized T-scores relative to a population mean of 50 and SD of 10, with a minimum of 15.4 and maximum of 73.3. Higher T-scores represent higher levels of physical function. Scores are calibrated against the general population.
Clinical Measure 9: Health-related quality of life assessed by the Patient Reported Outcomes Measurement Information System fatigue (v1.0) | Baseline and 10 weeks
  Patient Reported Outcomes Measurement Information System (PROMIS) are patient reported outcome surveys developed by the National Institutes for Health. This test is a computer adaptive test. Scores are represented as standardized T-scores relative to a population mean of 50 and SD of 10, with a minimum of 34.4 and maximum of 84.7. Higher T-scores represent higher levels of fatigue. Scores are calibrated against the general population.
Clinical Measure 10: Health-related quality of life assessed by the Patient Reported Outcomes Measurement Information System anxiety (v1.0) | Baseline and 10 weeks
  Patient Reported Outcomes Measurement Information System (PROMIS) are patient reported outcome surveys developed by the National Institutes for Health. This test is a computer adaptive test. Raw scores are converted to standardized T-scores relative to a population mean of 50 and SD of 10 (minimum T-score is 32.9, maximum is 84.9). Higher T-scores represent higher levels of anxiety. Scores are calibrated against the general population.
Clinical Measure 11: Health-related quality of life assessed by the Patient Reported Outcomes Measurement Information System depression (v1.0) | Baseline and 10 weeks
  Patient Reported Outcomes Measurement Information System (PROMIS) are patient reported outcome surveys developed by the National Institutes for Health. This test is a computer adaptive test. Scores are represented as standardized T-scores relative to a population mean of 50 and SD of 10 (minimum T-score is 34.2, maximum is 84.4). Higher T-scores represent higher levels of depression. Scores are calibrated against the general population.

CONTACTS AND LOCATIONS:
Overall Officials: Angela Senders, ND, MCR, Principal Investigator — Research Investigator and Assistant Professor
Locations (1):
- National University of Natural Medicine, Helfgott Research Institute, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li F, Harmer P, Fitzgerald K, Eckstrom E, Stock R, Galver J, Maddalozzo G, Batya SS. Tai chi and postural stability in patients with Parkinson's disease. N Engl J Med. 2012 Feb 9;366(6):511-9. doi: 10.1056/NEJMoa1107911. PMID 22316445
- [Background] Amano S, Nocera JR, Vallabhajosula S, Juncos JL, Gregor RJ, Waddell DE, Wolf SL, Hass CJ. The effect of Tai Chi exercise on gait initiation and gait performance in persons with Parkinson's disease. Parkinsonism Relat Disord. 2013 Nov;19(11):955-60. doi: 10.1016/j.parkreldis.2013.06.007. Epub 2013 Jul 5. PMID 23835431
- [Background] Schmitz-Hubsch T, Pyfer D, Kielwein K, Fimmers R, Klockgether T, Wullner U. Qigong exercise for the symptoms of Parkinson's disease: a randomized, controlled pilot study. Mov Disord. 2006 Apr;21(4):543-8. doi: 10.1002/mds.20705. PMID 16229022
- [Background] Wayne PM, Buring JE, Davis RB, Connors EM, Bonato P, Patritti B, Fischer M, Yeh GY, Cohen CJ, Carroll D, Kiel DP. Tai Chi for osteopenic women: design and rationale of a pragmatic randomized controlled trial. BMC Musculoskelet Disord. 2010 Mar 1;11:40. doi: 10.1186/1471-2474-11-40. PMID 20193083
- [Background] D'Souza E. Modified Fatigue Impact Scale - 5-item version (MFIS-5). Occup Med (Lond). 2016 Apr;66(3):256-7. doi: 10.1093/occmed/kqv106. No abstract available. PMID 27016749
- [Background] Hobart JC, Riazi A, Lamping DL, Fitzpatrick R, Thompson AJ. Measuring the impact of MS on walking ability: the 12-Item MS Walking Scale (MSWS-12). Neurology. 2003 Jan 14;60(1):31-6. doi: 10.1212/wnl.60.1.31. PMID 12525714
- [Background] Hobart J, Lamping D, Fitzpatrick R, Riazi A, Thompson A. The Multiple Sclerosis Impact Scale (MSIS-29): a new patient-based outcome measure. Brain. 2001 May;124(Pt 5):962-73. doi: 10.1093/brain/124.5.962. PMID 11335698
- [Background] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946
- [Background] Learmonth YC, Dlugonski DD, Pilutti LA, Sandroff BM, Motl RW. The reliability, precision and clinically meaningful change of walking assessments in multiple sclerosis. Mult Scler. 2013 Nov;19(13):1784-91. doi: 10.1177/1352458513483890. Epub 2013 Apr 15. PMID 23587605
- [Background] Chan JS, Ho RT, Wang CW, Yuen LP, Sham JS, Chan CL. Effects of qigong exercise on fatigue, anxiety, and depressive symptoms of patients with chronic fatigue syndrome-like illness: a randomized controlled trial. Evid Based Complement Alternat Med. 2013;2013:485341. doi: 10.1155/2013/485341. Epub 2013 Jul 31. PMID 23983785
- [Background] Ni X, Liu S, Lu F, Shi X, Guo X. Efficacy and safety of Tai Chi for Parkinson's disease: a systematic review and meta-analysis of randomized controlled trials. PLoS One. 2014 Jun 13;9(6):e99377. doi: 10.1371/journal.pone.0099377. eCollection 2014. PMID 24927169
- [Background] Ho RT, Chan JS, Wang CW, Lau BW, So KF, Yuen LP, Sham JS, Chan CL. A randomized controlled trial of qigong exercise on fatigue symptoms, functioning, and telomerase activity in persons with chronic fatigue or chronic fatigue syndrome. Ann Behav Med. 2012 Oct;44(2):160-70. doi: 10.1007/s12160-012-9381-6. PMID 22736201
- [Background] Oh B, Butow P, Mullan B, Clarke S, Beale P, Pavlakis N, Kothe E, Lam L, Rosenthal D. Impact of medical Qigong on quality of life, fatigue, mood and inflammation in cancer patients: a randomized controlled trial. Ann Oncol. 2010 Mar;21(3):608-614. doi: 10.1093/annonc/mdp479. Epub 2009 Oct 30. PMID 19880433
- [Background] Mills N, Allen J. Mindfulness of movement as a coping strategy in multiple sclerosis. A pilot study. Gen Hosp Psychiatry. 2000 Nov-Dec;22(6):425-31. doi: 10.1016/s0163-8343(00)00100-6. PMID 11072058
- [Background] Asano M, Finlayson ML. Meta-analysis of three different types of fatigue management interventions for people with multiple sclerosis: exercise, education, and medication. Mult Scler Int. 2014;2014:798285. doi: 10.1155/2014/798285. Epub 2014 May 14. PMID 24963407
- [Background] Beckerman H, Blikman LJ, Heine M, Malekzadeh A, Teunissen CE, Bussmann JB, Kwakkel G, van Meeteren J, de Groot V; TREFAMS-ACE study group. The effectiveness of aerobic training, cognitive behavioural therapy, and energy conservation management in treating MS-related fatigue: the design of the TREFAMS-ACE programme. Trials. 2013 Aug 12;14:250. doi: 10.1186/1745-6215-14-250. PMID 23938046
- [Background] Carter AM, Daley AJ, Kesterton SW, Woodroofe NM, Saxton JM, Sharrack B. Pragmatic exercise intervention in people with mild to moderate multiple sclerosis: a randomised controlled feasibility study. Contemp Clin Trials. 2013 Jul;35(2):40-7. doi: 10.1016/j.cct.2013.04.003. Epub 2013 Apr 21. PMID 23612222
- [Background] Ensari I, Motl RW, Pilutti LA. Exercise training improves depressive symptoms in people with multiple sclerosis: results of a meta-analysis. J Psychosom Res. 2014 Jun;76(6):465-71. doi: 10.1016/j.jpsychores.2014.03.014. Epub 2014 Mar 31. PMID 24840141
- [Background] Latimer-Cheung AE, Pilutti LA, Hicks AL, Martin Ginis KA, Fenuta AM, MacKibbon KA, Motl RW. Effects of exercise training on fitness, mobility, fatigue, and health-related quality of life among adults with multiple sclerosis: a systematic review to inform guideline development. Arch Phys Med Rehabil. 2013 Sep;94(9):1800-1828.e3. doi: 10.1016/j.apmr.2013.04.020. Epub 2013 May 10. PMID 23669008
- [Background] Marck CH, Hadgkiss EJ, Weiland TJ, van der Meer DM, Pereira NG, Jelinek GA. Physical activity and associated levels of disability and quality of life in people with multiple sclerosis: a large international survey. BMC Neurol. 2014 Jul 12;14:143. doi: 10.1186/1471-2377-14-143. PMID 25016312
- [Background] Mayo NE, Bayley M, Duquette P, Lapierre Y, Anderson R, Bartlett S. The role of exercise in modifying outcomes for people with multiple sclerosis: a randomized trial. BMC Neurol. 2013 Jun 28;13:69. doi: 10.1186/1471-2377-13-69. PMID 23809312
- [Background] Pilutti LA, Dlugonski D, Sandroff BM, Klaren R, Motl RW. Randomized controlled trial of a behavioral intervention targeting symptoms and physical activity in multiple sclerosis. Mult Scler. 2014 Apr;20(5):594-601. doi: 10.1177/1352458513503391. Epub 2013 Sep 5. PMID 24009162
- [Background] Guo LY, Yang CP, You YL, Chen SK, Yang CH, Hou YY, Wu WL. Underlying mechanisms of Tai-Chi-Chuan training for improving balance ability in the elders. Chin J Integr Med. 2014 Jun;20(6):409-15. doi: 10.1007/s11655-013-1533-4. Epub 2014 Jun 21. PMID 24952168
- [Background] Gonzalez Lopez-Arza MV, Varela-Donoso E, Montanero-Fernandez J, Rodriguez-Mansilla J, Gonzalez-Sanchez B, Gonzalez Lopez-Arza L. Qigong improves balance in young women: a pilot study. J Integr Med. 2013 Jul;11(4):241-5. doi: 10.3736/jintegrmed2013038. PMID 23867242
- [Background] Wu CY, Han HM, Huang MC, Chen YM, Yu WP, Weng LC. Effect of qigong training on fatigue in haemodialysis patients: A non-randomized controlled trial. Complement Ther Med. 2014 Apr;22(2):244-50. doi: 10.1016/j.ctim.2014.01.004. Epub 2014 Jan 10. PMID 24731895
- [Background] Sawynok J, Lynch M, Marcon D. Extension trial of qigong for fibromyalgia: a quantitative and qualitative study. Evid Based Complement Alternat Med. 2013;2013:726062. doi: 10.1155/2013/726062. Epub 2013 Aug 28. PMID 24069054
- [Background] Haak T, Scott B. The effect of Qigong on fibromyalgia (FMS): a controlled randomized study. Disabil Rehabil. 2008;30(8):625-33. doi: 10.1080/09638280701400540. PMID 17852292
- [Background] Warner L, McNeill ME. Mental imagery and its potential for physical therapy. Phys Ther. 1988 Apr;68(4):516-21. doi: 10.1093/ptj/68.4.516. PMID 3281175
- [Background] Paul L, Coote S, Crosbie J, Dixon D, Hale L, Holloway E, McCrone P, Miller L, Saxton J, Sincock C, White L. Core outcome measures for exercise studies in people with multiple sclerosis: recommendations from a multidisciplinary consensus meeting. Mult Scler. 2014 Oct;20(12):1641-50. doi: 10.1177/1352458514526944. Epub 2014 Mar 17. PMID 24639480
- [Background] Senders A, Hanes D, Bourdette D, Whitham R, Shinto L. Reducing survey burden: feasibility and validity of PROMIS measures in multiple sclerosis. Mult Scler. 2014 Jul;20(8):1102-11. doi: 10.1177/1352458513517279. Epub 2014 Jan 8. PMID 24402035
- [Background] Fisk JD, Ritvo PG, Ross L, Haase DA, Marrie TJ, Schlech WF. Measuring the functional impact of fatigue: initial validation of the fatigue impact scale. Clin Infect Dis. 1994 Jan;18 Suppl 1:S79-83. doi: 10.1093/clinids/18.supplement_1.s79. PMID 8148458
- [Background] Dite W, Temple VA. A clinical test of stepping and change of direction to identify multiple falling older adults. Arch Phys Med Rehabil. 2002 Nov;83(11):1566-71. doi: 10.1053/apmr.2002.35469. PMID 12422327
- [Background] Linke SE, Gallo LC, Norman GJ. Attrition and adherence rates of sustained vs. intermittent exercise interventions. Ann Behav Med. 2011 Oct;42(2):197-209. doi: 10.1007/s12160-011-9279-8. PMID 21604068
- [Background] Yost KJ, Eton DT, Garcia SF, Cella D. Minimally important differences were estimated for six Patient-Reported Outcomes Measurement Information System-Cancer scales in advanced-stage cancer patients. J Clin Epidemiol. 2011 May;64(5):507-16. doi: 10.1016/j.jclinepi.2010.11.018. PMID 21447427
- [Result] Ben-Zacharia AB. Therapeutics for multiple sclerosis symptoms. Mt Sinai J Med. 2011 Mar-Apr;78(2):176-91. doi: 10.1002/msj.20245. PMID 21425263
- [Result] Nilsagard Y, Gunn H, Freeman J, Hoang P, Lord S, Mazumder R, Cameron M. Falls in people with MS--an individual data meta-analysis from studies from Australia, Sweden, United Kingdom and the United States. Mult Scler. 2015 Jan;21(1):92-100. doi: 10.1177/1352458514538884. Epub 2014 Jun 16. PMID 24948687
- [Result] Peterson EW, Cho CC, von Koch L, Finlayson ML. Injurious falls among middle aged and older adults with multiple sclerosis. Arch Phys Med Rehabil. 2008 Jun;89(6):1031-7. doi: 10.1016/j.apmr.2007.10.043. PMID 18503796
- [Result] Fischer M, Fugate-Woods N, Wayne PM. Use of pragmatic community-based interventions to enhance recruitment and adherence in a randomized trial of Tai Chi for women with osteopenia: insights from a qualitative substudy. Menopause. 2014 Nov;21(11):1181-9. doi: 10.1097/GME.0000000000000257. PMID 24845395
- [Result] Motl RW, Cohen JA, Benedict R, Phillips G, LaRocca N, Hudson LD, Rudick R; Multiple Sclerosis Outcome Assessments Consortium. Validity of the timed 25-foot walk as an ambulatory performance outcome measure for multiple sclerosis. Mult Scler. 2017 Apr;23(5):704-710. doi: 10.1177/1352458517690823. Epub 2017 Feb 16. PMID 28206828
- [Result] Taylor E, Taylor-Piliae RE. The effects of Tai Chi on physical and psychosocial function among persons with multiple sclerosis: A systematic review. Complement Ther Med. 2017 Apr;31:100-108. doi: 10.1016/j.ctim.2017.03.001. Epub 2017 Mar 2. PMID 28434462
- [Derived] Buttolph L, Wooliscroft L, Bradley R, Zwickey H. Participant Perspectives on Community Qigong for People with Multiple Sclerosis. Integr Med Rep. 2023 Feb 1;2(1):26-34. doi: 10.1089/imr.2022.0079. Epub 2023 Feb 1. PMID 36895618
- [Derived] Buttolph L, Corn J, Hanes D, Bradley R, Senders A. Community qigong for People with Multiple Sclerosis: A Pragmatic Feasibility Study. J Altern Complement Med. 2021 Jun;27(6):506-514. doi: 10.1089/acm.2020.0481. Epub 2021 Mar 26. PMID 33769837
- See also: Definition of Multiple Sclerosis — https://www.nationalmssociety.org/What-is-MS/Definition-of-MS

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-10-06): https://cdn.clinicaltrials.gov/large-docs/59/NCT04585659/Prot_SAP_000.pdf
  • Informed Consent Form (2016-10-06): https://cdn.clinicaltrials.gov/large-docs/59/NCT04585659/ICF_001.pdf